CLINICAL TRIAL: NCT03219346
Title: The Effectiveness of Oral Health in Improving Dysphagia of Patients After Stroke of Swallowing Function and Oral Health Quality of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsiao-Jung Chen, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201700143B0
Record Dates: First submitted 2017-07-11; First posted 2017-07-17 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Swallowing Disorders; Stroke
Keywords: stroke , swallowing function ,oral health quality of life
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral hygiene (Experimental)
  Interventions: Other: oral care program

INTERVENTIONS:
Other: oral care program — Oral care (sputum and special needs of people cleaning teeth) time for three days a week (with swallowing treatment time before), once a day, each about 10 minutes of oral care program.

SUMMARY:
The prevalence of chewing dysphagia in the domestic rehabilitation department ward was about 53.61%.Nasal tube retention of about 31%, due to nasogastric tube feeding, often overlooked oral hygiene, easy to cause respiratory tract infection. At the same time, oral hygiene will also affect the effectiveness of swallowing treatment, is worthy of attention to health problems.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of first stroke with nasal tube retention
2. Language therapist providing swallowing treatment
3. Caregiver providing oral care to patients

Exclusion Criteria:

1. Oral cancer
2. head and neck cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-02-10 (Estimated); Study Completion 2019-02-17 (Estimated)

PRIMARY OUTCOMES:
Functional oral intake scale | before the first swallowing treatment (one day before treatment)
  Seven different grades,Normal for 7 points;Total score of 1-7

SECONDARY OUTCOMES:
Functional oral intake scale | two weeks after the swallowing treatment (14 days)
  Seven different grades,Normal for 7 points;Total score of 1-7
Functional oral intake scale | three weeks after the swallowing treatment (21 days)
  Seven different grades,Normal for 7 points;Total score of 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Ting Hung, Study Director — Chang Gung University
Locations (1):
- Chang Gung University, Taipei, Taiwan